CLINICAL TRIAL: NCT04984096
Title: Treatment Patterns and Clinical Outcomes Among Patients Receiving Anlotinib in Combination With PD-1 Inhibitor for Advanced/Metastatic Esophageal Squamous Cell Carcinoma in Real-world Settings(APEC)
Brief Title: Anlotinib Combined With PD-1 Inhibitors for Advanced/Metastatic Esophageal Cancer
Acronym: APEC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jun Liu, associate proffessor, Shanghai Chest Hospital
Other Study IDs: ShanghaiChest RT
Record Dates: First submitted 2021-07-24; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Efficacy and Safety of Anlotinib combined with PD-1 inhibitors as 2 or more lines treatment for Heavily Pretreated Patients With Advanced, Metastatic Squamous Cell Carcinoma of the Esophagus.

DETAILED DESCRIPTION:
The APEC study is a multi-center, retrospective ,real-world study of anlotinib combined with PD-1 inhibitors for patients with histologically confirmed advanced and metastatic esophageal squamous cell carcinoma (ESCC) that progressed after 1or more lines of therapy, conducted at 8 sites in China. Patients received anlotinib combined with PD-1 inhibitors , every 3 weeks for up to 2 years, until progression of disease, unacceptable toxic effects occurred, or withdrawal of consent. The primary end point was the progression-free survival (PFS)among all patients. Secondary end points included Adverse events (AEs),objective response rate (ORR) ,duration of response (DOR), , and overall survival (OS). Tumor response was assessed per the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged more than 18 years old;
2. ECOG PS：0-2;
3. Subjects with histologically or cytologically confirmed locally advanced and/or advanced esophageal squamous cell carcinoma(ESCC);
4. For local advanced or advanced ESCC, disease progression occurred after 1 or more lines systemic treatment previously;
5. Have received anlotinib combined with PD-1 inhibitor treatment.

Exclusion Criteria:

1. have used Anlotinib before;
2. mixed with small cell cancer and/or other kinds of cancer ;
3. Previously (within 5 years) or presently suffering from other malignancies;
4. Symptomatic or uncontrolled brain metastases;
5. Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months or serious cardiac arrhythmia requiring medication;
6. Pregnancy or lactation. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal squamous cell carcinoma who have received anlotinib combined with PD-1 inhibitors as 2 or more lines treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months
  PFS is defined as the time from the date of treatment to the first date of disease progression or death from any cause

SECONDARY OUTCOMES:
Adverse Events | Until 30 day safety follow-up visit
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 12 months)
  Treatment response are defined as complete response (CR), partial response (PR), stable disease (SD) and progression disease (PD) according to Response Evaluation Criteria in Solid Tumor (RECISIT criteria, version 1.1) and the percentage of patients who achieved CR, PR and SD was defined as disease control rate (DCR).
Overall Survival (OS) | 12 months
  OS is calculated from diagnosis to death or last follow-up time

REFERENCES:
- [Derived] Zhu X, Ma X, Li H, Zhang M, Cheng Y, Wu J, Yu W, Feng W, Zhao L, Li Z, Fu X, Liu J. The efficacy and safety of anlotinib plus PD-1 inhibitor in locally advanced/metastatic esophageal squamous cell carcinoma (ESCC) patients who progressed on prior immune checkpoint inhibitors (ICIs): a retrospective real-world study (NCT 04984096). Ann Med. 2025 Dec;57(1):2443811. doi: 10.1080/07853890.2024.2443811. Epub 2024 Dec 23. PMID 39711430